CLINICAL TRIAL: NCT02594436
Title: The Use of Picato® (Ingenol Mebutate) to Treat Actinic Keratosis in Standard Clinical Practice: A Prospective Phase IV, Multicentre, Pan-Hellenic Observational Cohort Study
Brief Title: The Use of Picato® (Ingenol Mebutate) to Treat Actinic Keratosis in Standard Clinical Practice
Acronym: PrAKtice
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PICATO-1220
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; topical; ingenol mebutate; Picato®
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ingenol mebutate gel 0.015 percent: Topical treatment of face or scalp once daily for three consecutive days
  Interventions: Drug: Ingenol mebutate
- Ingenol mebutate gel 0.05 percent: Topical treatment of trunk or extremities once daily for two consecutive days
  Interventions: Drug: Ingenol mebutate

INTERVENTIONS:
Drug: Ingenol mebutate — Non-Interventional study enrolling patients already planned to be treated with ingenol mebutate according to approved labelling
  Other Names: Picato

SUMMARY:
This is a prospective, non-interventional study of adult patients prescribed topical treatment with ingenol mebutate gel (Picato®) as part of provision of care for the treatment of Non-hyperkeratotic, non-hypertrophic Actinic Keratosis (AK). Patients with complete clearance at 8 weeks will be followed for one year or until retreatment of AK in the area initially treated, whatever comes first. For patients with incomplete clearance in the treated area at 8 weeks the treatment strategy for this area will be recorded but no further follow-up will take place. The effectiveness, tolerability, adherence, patient satisfaction and health-related quality of life (HRQoL) associated with Picato® treatment will be evaluated.

DETAILED DESCRIPTION:
Actinic Keratosis (AK) is caused by exposure to UV radiation and has the potential to regress to normal skin or to progress to squamous cell carcinoma. Ingenol mebutate gel is a relatively new topical treatment option for AK in Greece.

Taking into consideration the limited real-world evidence that is attributed to the recent advent of Picato in the Greek market, this non-interventional observational study aims primarily at assessing the characteristics of patients selected for this treatment, the effectiveness and tolerability of the treatment, patient satisfaction and the impact of the therapy on patients' HRQoL in standard clinical practice.The study will be carried out by approximately 30 physicians practicing in private or public hospitals and clinics in representative geographical regions of Greece.

ELIGIBILITY:
Inclusion Criteria:

* Planned to receive topical ingenol mebutate gel for treatment of Actinic Keratosis according to current labelling in Greece.
* Written informed consent obtained to use the patient's data for the study.

Exclusion Criteria:

* Contraindications according to prescribing information.
* Previous treatment with PICATO in the selected treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients planned for starting treatment non-hyperkeratotic, non-hypertrophic actinic keratosis on face, scalp, trunk or extremities with topical ingenol mebutate gel.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Rate of complete clearance | Around 8 weeks post treatment
  Percentage of patients with no clinically visible remaining lesions in treated area
Lesion count reduction | Around 8 weeks post treatment
  Reduction in number of clinically visible lesions in treated area compared to baseline count.

SECONDARY OUTCOMES:
Remission rate for patients with complete initial clearance | 12 months
  Proportion of patients without known recurrence of AK lesions in treated area for patients with complete initial clearance
Patient satisfaction with treatment | Around 8 weeks post treatment
  Patient reported satisfaction with treatment as measured by the domains of effectiveness, convenience and global satisfaction of TSQM-9 (Treatment Satisfaction Questionnaire of Medication)
Health Related Quality of Life EQ-5D-5L | Baseline and around 8 weeks post treatment
  EQ-5D-5L is a standardized instrument for use as a measure of health outcome. It provides a simple descriptive profile and a single index value for health status. EQ-5D-5L is designed for self-completion by respondents. It consists of two pages comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Sitaras, MD, Study Director — LEO Pharma Hellas SA
Locations (1):
- Office Based Physician, Athens, Peristeri, Greece